CLINICAL TRIAL: NCT07270055
Title: Effect of Neonatal Device Swaddy® on the Stress Level of Preterm Newborns: A Randomized Clinical Trial.
Brief Title: Swaddy, a Neonatal Positioning Device.
Acronym: Swaddy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Fundació Institut Germans Trias i Pujol (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IIBSP-SWA-2025-35
Record Dates: First submitted 2025-11-14; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Stress

STUDY DESIGN:
Intervention Model Description: Randomized, crossover, multicenter, open-label clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Swaddy first (Active Comparator): In this project, patients will be randomized into two groups. In Group 1, on the first day (day 1), the first measurement (baseline) will be made. Subsequently, the Swaddy® containment device will be placed and the containment will be maintained for 3 hours, in which the same variables will be measured: Heart Rate (HR), Respiratory Rate (RF), temperature, O2 Saturation (SatO2) and pain scale at 60, 120 and 180 minutes. This procedure will be repeated on day 2 and 3. On day 4, the same measurements will be carried out using standard containment care. This procedure will be repeated on days 5 and 6 (all three at approximately the same time of day as in the intervention).
  Interventions: Device: Swaddy day 1, 2, 3
- Group Swaddy second (Active Comparator): In Group 2, on the first day (day 1), the first measurement (baseline) will be taken. Subsequently, the patient will be kept in an incubator for 3 hours, in which the following variables will be measured: Heart Rate (HR), Respiratory Rate (RF), temperature, O2 Saturation (SatO2) and pain scale at 60, 120 and 180 minutes, using standard containment care. This procedure will be repeated on day 2 and 3. On day 4, the same measurements will be carried out by applying containment with the Swaddy® device and will be repeated on days 5 and 6.
  Interventions: Device: Swaddy day 4, 5, 6

INTERVENTIONS:
Device: Swaddy day 1, 2, 3 — In Group 1, on the first day (day 1), the first measurement (baseline) will be made. Subsequently, the Swaddy® containment device will be placed and the containment will be maintained for 3 hours, in which the same variables will be measured: Heart Rate (HR), Respiratory Rate (RF), temperature, O2 Saturation (SatO2) and pain scale at 60, 120 and 180 minutes. This procedure will be repeated on day 2 and 3. On day 4, the same measurements will be carried out using standard containment care. This procedure will be repeated on days 5 and 6 (all three at approximately the same time of day as in the intervention).
  Arms: Group Swaddy first
Device: Swaddy day 4, 5, 6 — In Group 2, on the first day (day 1), the first measurement (baseline) will be taken. Subsequently, the patient will be kept in an incubator for 3 hours, in which the following variables will be measured: Heart Rate (HR), Respiratory Rate (RF), temperature, O2 Saturation (SatO2) and pain scale at 60, 120 and 180 minutes, using standard containment care. This procedure will be repeated on day 2 and 3. On day 4, the same measurements will be carried out by applying containment with the Swaddy® device and will be repeated on days 5 and 6.
  Arms: Group Swaddy second

SUMMARY:
The objective of this clinical trial is to evaluate the effect of positional restraint on the stress level of preterm newborns, resting in the incubator. The main question sought to be answered is: The stress level of the preterm newborn will decrease with swaddy® containment, compared to standard care, and both with similar safety.

Participants will remain in the incubator for 3 consecutive hours and the level of stress in the same patient will be evaluated, one day with containment and another day without containment.

DETAILED DESCRIPTION:
Primary objective: To assess the effect of Swaddy® containment on the stress level of newborns ≤1500 grams at birth admitted to a NICU, using the Comfort B Scale, for a maximum period of 3 consecutive hours, compared to standard containment care.

Secondary objectives:

* To evaluate the effect of positional restraint with Swaddy® on the stability of the preterm newborn, through the physiological parameters HR, RF, temperature, and SatO2, compared to standard containment care for 3 consecutive hours.
* To evaluate the safety of the number of apneas, in containment with Swaddy® compared to standard care.

Swaddy®, is an adjustable garment of clothing, with a built-in cap, which favors the symmetry of limbs with midline of the body and the hand-to-hand and hand-to-mouth position of preterm newborns, very conciliatory positions for these patients. Its fabric is thin and soft, to prevent overheating, and elastic, to favor the flexor position and allow some mobility. It is a device designed by the IP of the project, registered and patented by the Institut de Recerca Sant Pau, and currently marketed.

In this project, patients will be randomized into two groups. In Group 1, on the first day (day 1), the first measurement (baseline) will be made. Subsequently, the Swaddy® containment device will be placed and the containment will be maintained for 3 hours, in which the same variables will be measured: Heart Rate (HR), Respiratory Rate (RF), temperature, O2 Saturation (SatO2) and pain scale at 60, 120 and 180 minutes. This procedure will be repeated on day 2 and 3. On day 4, the same measurements will be carried out using standard containment care. This procedure will be repeated on days 5 and 6 (all three at approximately the same time of day as in the intervention). In Group 2, it will be done in reverse.

Vital signs HR, RF, oxygen saturation will be measured with the patient's monitor and temperature with a skin sensor in the incubator itself, which will be located in the patient's thoracoabdominal area.

To assess the safety of the device, the number of apneas of prematurity performed with Swaddy® containment and standard care will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Newborns weighing ≤1500 grams at birth admitted to the NICU. • Patients who are in an incubator.

Exclusion Criteria:

* Hemodynamic instability.

  * Be a carrier of CPAP or nasal BIPAP with a cap (because the CPAP/BIPAP already has a built-in cap, just like Swaddy).
  * Be in treatment with phototherapy.

Min Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Comfort B scale | three hours during the intervention
  It is a scale validated in pediatrics that assesses the behavioral signs of the newborn. Its maximum value is 30 and its minimum is 6. And the higher score, is the greater the pain or stress.

SECONDARY OUTCOMES:
Heart rate | three hours during the intervention
  Heart rate
Respiratory rate | three hours during the intervention
  Respiratory rate
Oxygen saturation | three hours during the intervention
  Oxygen saturation
Temperature | three hours during the intervention
  Temperature

IPD SHARING:
Plan to Share IPD: No